CLINICAL TRIAL: NCT03515668
Title: The Influence of Dopamine Activity on Neuromuscular Function During Passive Heat Stress
Brief Title: Dopamine and Muscle Function in the Heat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, Stephen Cheung, Professor, Brock University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 17-123
Record Dates: First submitted 2018-04-23; First posted 2018-05-03 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Muscle Force; Hyperthermia
MeSH Terms: conditions — Hyperthermia | interventions — Methylphenidate; Tablets

STUDY DESIGN:
Intervention Model Description: Healthy males 18-30 years of age
Who Masked: Investigator
Masking Description: Double-blinding of participant and investigator, with independent investigator in charge of placebo and drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ritalin (Experimental): 20 mg Ritalin, 90 min before testing
  Interventions: Drug: Ritalin 20 mg Tablet
- Control (Placebo Comparator): Identical size/taste placebo pill, 90 min before testing
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Ritalin 20 mg Tablet — Single dose for all participants
  Arms: Ritalin
Drug: Placebo Oral Tablet — Placebo with same appearance/taste
  Arms: Control

SUMMARY:
our goal is to study the effects of dopamine activity, using Ritalin ingestion, on neuromuscular function over the course of a progressive heating and cooling protocol developed in our lab. We hypothesize that Ritalin will minimize the previously reported progressive impairment in neuromuscular function with hyperthermia compared to placebo, suggesting that dopamine activity preserves neuromuscular capacity with hyperthermia.

DETAILED DESCRIPTION:
Increased core temperature (hyperthermia) has been associated with impaired neuromuscular performance, with the majority of research suggesting that the observed fatigue is related to the central nervous system. Small doses of Ritalin has been used to study how changes in dopamine activity affects exercise capacity in the heat. This study found that 20 mg of Ritalin had no effect on exercise capacity in a thermoneutral environment of 18°C. However, when in a hot (30°C) environment, the Ritalin resulted in a 16% improvement in finishing time compared to the placebo trial. Interestingly, the higher output during the Ritalin-hot condition also resulted in higher rates of heat production and a higher (~0.6°C) core temperature, suggesting that dopamine enabled greater voluntary tolerance of hyperthermia. This matches recent work from our own work showing that motivational skills training increased both exercise tolerance and final core temperature, and it is possible that dopamine activity played a role in this improvement.

Ultimately, fatigue is shown in an inability to sustain muscular force. However, the role of dopamine activity on neuromuscular function (e.g., central activation and recruitment of muscle) during hyperthermia is unknown. One study reported that 20 mg of Ritalin did not alter neuromuscular function, but this study was done without thermal stress.

Therefore, our goal is to study the effects of dopamine activity, using Ritalin ingestion, on neuromuscular function over the course of a progressive heating and cooling protocol developed in our lab. We hypothesize that Ritalin will minimize the previously reported progressive impairment in neuromuscular function with hyperthermia (5, 7) compared to placebo, suggesting that dopamine activity preserves neuromuscular capacity with hyperthermia.

ELIGIBILITY:
Inclusion Criteria:

* High aerobic fitness (>55 mL/kg/min maximal aerobic capacity)

Exclusion Criteria:

* diagnosed cardiovascular, respiratory and/or neuromuscular disease, prescription of Ritalin or any drugs for hyperactivity within the past 1 year, any current prescription medication (except for asthma/allergy inhalers), any contraindications to Ritalin.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Wrist flexion torque | 2-4 hours after ingestion
  Maximal voluntary contraction of wrist flexion

CONTACTS AND LOCATIONS:
Locations (1):
- Brock University, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No sharing planned